CLINICAL TRIAL: NCT03361605
Title: Neuroimaging of Anesthetic Modulation of Human Consciousness
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Anthony G Hudetz, Professor of Anesthesiology, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00103361
Record Dates: First submitted 2017-11-03; First posted 2017-12-05 (Actual); Results first posted 2020-08-05 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Healthy
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Propofol Administration (Experimental)
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Propofol administration

SUMMARY:
This study's purpose is to see if mental functions take place during different levels of anesthesia, using a commonly used drug (Propofol). fMRI (functional Magnetic Resonance Imaging, or "brain imaging") shows areas in the brain involved in thinking at different depths of anesthesia.

DETAILED DESCRIPTION:
Administering anesthetic drugs to suppress consciousness is an imperatively important step in major surgical operations. Yet the neurobiological mechanisms that underlie loss of consciousness under general anesthesia remain elusive. Despite advancements in understanding the molecular, synaptic, and cellular effects of anesthetics, the large-scale, systems-level modulation of neuronal processes that support conscious cognitive functions is incompletely understood. While profound decreases in global and regional brain metabolism, blood flow, and functional connectivity have been reported, these changes often fail to correlate with the loss and return of consciousness. To date, there is no "consciousness meter" or "gold standard" to objectively assess and monitor the level of consciousness under general anesthesia. Several studies suggest that residual cognitive functions may not completely vanish under general anesthesia; however, the level and complexity of residual information processing in the anesthetized brain remains unknown. Finally, the neurobiological mechanisms that govern anesthesia induction and emergence appear to be partially different, but the relevance of these differences to the modulation of the state of consciousness is unclear.

ELIGIBILITY:
Inclusion Criteria:

1. Must have a body mass index (BMI) less than 30.
2. Must be right handed
3. Must be English speaking
4. Must be capable of giving written informed consent.
5. Must have history of playing tennis (or any type of racquet sport) at least 30 times over lifetime.

Exclusion Criteria:

1. History of obstructive sleep apnea;
2. History of a difficult airway with a previous anesthetic;
3. History of neurological disorders;
4. Hypertension or other cardiovascular abnormalities;
5. Pulmonary hypertension or other pulmonary abnormalities;
6. Gastroesophageal reflux disease (GERD) or heartburn;
7. History of significant head injury with loss of consciousness;
8. Learning disability or other developmental disorder;
9. Allergic reactions to eggs;
10. Pregnant or nursing mothers;
11. Contraindications to neuroimaging methods;
12. Inability or unwilling to fast, or withhold food and liquid intake, for 8 hours prior to your scheduled study visit.
13. Unwilling to abstain from alcohol use for 24 hours prior to your scheduled study visit.
14. History of drug use, or have a positive drug screen.
15. Tattoos on the head or neck region - all other tattoos are subject to determination by investigators.
16. Any impairment, activity or situation that in the judgment of the study coordinator or Principal Investigators would prevent satisfactory completion of the study protocol.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony G Hudetz, PhD, Principal Investigator — University of Michigan
Locations (1):
- Michigan Medicine - University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Propofol Administration
Started | 29
Completed | 26
Not Completed | 3
Not completed — Analyzable data not available | 3

BASELINE CHARACTERISTICS:
Population: 29 participants were consented and received study drug.
Arm/Group | Propofol Administration
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 18
  More than one race | 0
  Unknown or Not Reported | 1
BOLD response [Mean (Standard Deviation); unit: percentage of BOLD signal change] — The BOLD (blood oxygen level-dependent) signal is the measured variable as obtained by functional magnetic resonance imaging (fMRI). It is an indirect, relative measure of local neuronal activity in the brain. Higher BOLD signal value indicates more neuronal activity. Population: Analyzable data was not available for four subjects
  percentage of BOLD signal change
    number analyzed (Participants) | 26
    (all) | 0.599 (0.244)
Squeeze pressure [Mean (Standard Deviation); unit: mmHg] — Population: Analyzable data was not available for four subjects
  mmHg
    number analyzed (Participants) | 26
    (all) | 13.98 (5.27)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Blood Oxygen Level Dependent (BOLD) Response to Sensory Stimuli During Sedation
Description: Change = BOLD Response During Sedation - BOLD Response During Baseline
Time Frame: Baseline to 90 minutes
Population: Intent to study brain activity change (BOLD response) during propofol administration
Measure: Mean (Standard Deviation); unit: percentage of BOLD signal change
Arm/Group | Propofol Administration
Number analyzed (Participants) | 26
percentage of BOLD signal change | -0.349 (0.223)
Statistical Analysis 1: Comparison: Propofol Administration; The null hypothesis is no difference in BOLD response between sedated state and baseline; Test type: Superiority — Our study adopted a within-subject design, which is not a randomized controlled trial (RCT) such as testing if one treatment is superior to another. Therefore, here the "Superiority" indicates if propofol administration has a statistically significant impact on the brain activity in response to sensory stimuli; p < 0.0001, t-test, 2 sided — The threshold for statistical significance was p=0.05. The p-value was not adjusted for multiple comparisons, as only one comparison was performed; Mean Difference (Net) = -0.349, Standard Deviation 0.223 — Difference = BOLD Response During Sedation - BOLD Response During Baseline

2. Secondary Outcome: Change From Baseline in Squeeze Pressure
Description: Measurements of the force of participants' hand squeezing on a rubber ball in response to instructions. Change = Squeeze Pressure During Sedation - Squeeze Pressure During Baseline.
Time Frame: Baseline to 90 minutes
Population: Intent to study squeeze pressure change during propofol administration
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | Propofol Administration
Number analyzed (Participants) | 26
Millimeter of mercury (mmHg) | -2.16 (3.09)
Statistical Analysis 1: Comparison: Propofol Administration; The null hypothesis is no difference in squeeze pressure between sedated state and baseline; Test type: Superiority — Our study adopted a within-subject design, which is not a randomized controlled trial (RCT) such as testing if one treatment is superior to another. Therefore, here the "Superiority" indicates if propofol administration has a statistically significant impact on the squeeze pressure in response to verbal instructions; p = 0.00148, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -2.16, Standard Deviation 3.09 — Difference = Squeeze Pressure During Sedation - Squeeze Pressure During Baseline

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Propofol Administration
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-10): https://cdn.clinicaltrials.gov/large-docs/05/NCT03361605/Prot_SAP_000.pdf